CLINICAL TRIAL: NCT02358889
Title: A Phase 2 Randomized, Double-masked, Multicenter, Active-controlled Study Evaluating Administration of Repeated Intravitreal Doses of hI-con1™ in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: Study Evaluating Intravitreal hI-con1™ in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Acronym: EMERGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iconic Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IT-002
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Choroidal Neovascularization; Age-related Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — hI-con1; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- hI-con1 (Experimental): Patients will receive monthly intravitreal hI-con1 as monotherapy (plus sham injection) for the first 2 months followed by monthly treatment for 3 months, as needed, according to protocol criteria.
  Interventions: Biological: hI-con1; Other: Sham injection
- hI-con1 + ranibizumab (Experimental): Patients will receive monthly intravitreal hI-con1 in combination with intravitreal ranibizumab for the first 2 months followed by monthly treatment for 3 months, as needed, according to protocol criteria.
  Interventions: Biological: hI-con1; Biological: ranibizumab
- ranibizumab (Active Comparator): Patients will receive monthly intravitreal ranibizumab as monotherapy (plus sham injection) for the first 2 months followed by monthly treatment for 3 months, as needed, according to protocol criteria.
  Interventions: Biological: ranibizumab; Other: Sham injection

INTERVENTIONS:
Biological: hI-con1 — Intravitreal injection of hI-con1 0.3 mg
  Other Names: human Immuno-conjugate 1
  Arms: hI-con1; hI-con1 + ranibizumab
Biological: ranibizumab — Intravitreal injection of ranibizumab 0.5 mg
  Other Names: Lucentis®
  Arms: hI-con1 + ranibizumab; ranibizumab
Other: Sham injection — No injection is given, a needleless syringe is used to mimic an injection.
  Arms: hI-con1; ranibizumab

SUMMARY:
The purpose of this study is to evaluate the safety, biological activity and pharmacodynamic effect of repeated intravitreal doses of hI-con1 0.3 mg administered as monotherapy and in combination with ranibizumab 0.5 mg compared to ranibizumab 0.5 mg monotherapy in treating patients with choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any race at least 50 years of age
* Active primary Choroidal Neovascularization (CNV) secondary to Age-Related Macular Degeneration (AMD) in the study eye
* Best Corrected Visual Acuity (BCVA) of 70 to 24 letters (worse than 20/40 up to 20/320) in the study eye

Exclusion Criteria:

* Monocular patient or patient with a BCVA of 35 or fewer letters (20/200 or worse) in the better seeing eye
* Any prior treatment of CNV or advanced AMD in the study eye, except for dietary supplements or vitamins
* Any intraocular or ocular surface surgery (including cataract surgery and laser procedures) in the study eye within 3 months
* Vitrectomy in the study eye
* Hereditary or chronic hemorrhagic or coagulopathy conditions (i.e., hemophilia)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Burian, MD, Study Director — Iconic Therapeutics, Inc.
Locations (47):
- United States (47):
  - Phoenix, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Campbell, California
  - Glendale, California
  - Laguna Hills, California
  - Mountain View, California
  - Palm Desert, California
  - Palo Alto, California
  - San Francisco, California
  - Santa Ana, California
  - Golden, Colorado
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - Panama City, Florida
  - Sarasota, Florida
  - Stuart, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Jackson, Michigan
  - Royal Oak, Michigan
  - West Bloomfield, Michigan
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - Bloomfield, New Jersey
  - Brooklyn, New York
  - Hauppauge, New York
  - Syracuse, New York
  - Ashland, Oregon
  - Portland, Oregon
  - Huntingdon Valley, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Columbia, South Carolina
  - Kingsport, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah
  - Silverdale, Washington
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
Started | 30 | 30 | 28
Completed | 30 | 28 | 27
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab | Total
Number analyzed (Participants) | 30 | 30 | 28 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (10.65) | 78.4 (9.92) | 78.8 (7.19) | 77.1 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 17 | 53
  Male | 11 | 13 | 11 | 35
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 28 | 88

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Month 3
Description: Best corrected visual acuity (BCVA) was measured pre treatment prior to dilating eyes, using standard Early Treatment Diabetic Retinopathy Study (ETDRS) retro illuminated charts. The BCVA was recorded as the total letter score in each eye.
Time Frame: Baseline and Month 3
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 29 | 30 | 27
Letters | .3 (7.76) | 6.8 (8.21) | 7.6 (7.05)

2. Primary Outcome: Change From Baseline in Central Retinal Subfield Thickness (CST) in the Study Eye at Month 3
Description: Optical Coherence Tomography (OCT) imaging was performed pre treatment during visits in which study treatment was administered and to assess lesion characteristics for the study eye. and were evaluated by a central reading center for standardized grading.
Time Frame: Baseline and Month 3
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 29 | 30 | 27
Microns | 53.9 (17.01) | 66.3 (10.95) | 64.9 (27)

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye at Month 6
Description: as for outcome 1
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 29 | 30 | 27
Letters | -2.1 (8.05) | 8.4 (10.14) | 8.3 (9.10)

4. Secondary Outcome: Change From Baseline in CST in the Study Eye at Month 6
Description: Central Retinal Subfield Thickness (CST) as measured by Optical Coherence Tomography (OCT). The change from the baseline measurement was compared to the month 6 measurement.
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
Number analyzed (Participants) | 29 | 30 | 27
Microns | -35.7 (71.52) | -83.9 (71.52) | -91.4 (137.10)

ADVERSE EVENTS:
Arm/Group | hI-con1 | hI-con1 + Ranibizumab | Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/30 | 1/30 | 5/28
Other Adverse Events (participants affected / at risk) | 21/30 | 26/30 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hI-con1 (N=30) | hI-con1 + Ranibizumab (N=30) | Ranibizumab (N=28)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vertigo Positional (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hI-con1 (N=30) | hI-con1 + Ranibizumab (N=30) | Ranibizumab (N=28)
Conjunctival Haemorrhge (Eye disorders) | 4 (4) | 8 (8) | 4 (4)
Vitreous Floaters (Eye disorders) | 4 (4) | 4 (4) | 3 (3)
Eye Pain (Eye disorders) | 1 (1) | 7 (7) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 8 (8) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Vitreous Detachment (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Conjunctival Oedema (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Punctate Keratitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Increased Intraocular Pressure (Eye disorders) | 5 (5) | 2 (2) | 0 (0)
Abnormal Visual Acuity Test (Eye disorders) | 5 (5) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No